CLINICAL TRIAL: NCT05229913
Title: Effects of Different Concentrations of Esketamine on Postpartum Depression After Cesarean Section
Brief Title: Effects of Esketamine on Postpartum Depression
Acronym: EEPD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qinghai University (Other)
Collaborators: Qinghai Red Cross Hospital (Other)
Responsible Party: Principal Investigator, Yang Jingmei, Principal Investigator, Qinghai University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: JMYang; 2019-ZJ-930 (Other Grant/Funding Number: Wang Xuejun)
Record Dates: First submitted 2022-01-05; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Postpartum Depression
Keywords: Esketamine; Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- The control group （Esketamine is not added） (Placebo Comparator): Postoperative intravenous analgesia pump formula：Sufentanil 1ug/kg+ Flurbiprofen Axetil 200mg The intravenous analgesic pump in each group was supplemented with normal saline and matched to 100 ml, the background infusion rate is 2ml/h, the Self-controlled intravenous analgesia pressing once dose is 1ml, the locking time is 20min, and the analgesia lasted until 48h after surgery.
  Interventions: Drug: Esketamine is not added
- Esketamine experimental group(E0.2) (Experimental): Postoperative intravenous analgesia pump formula：Esketamine 0.2mg/kg + Sufentanil 1ug/kg+ Flurbiprofen Axetil 200mg The intravenous analgesic pump in each group was supplemented with normal saline and matched to 100 ml, the background infusion rate is 2ml/h, the Self-controlled intravenous analgesia pressing once dose is 1ml, the locking time is 20min, and the analgesia lasted until 48h after surgery.
  Interventions: Drug: Esketamine 0.2mg/kg
- Esketamine experimental group (E0.4) (Experimental): Postoperative intravenous analgesia pump formula：Esketamine 0.4mg/kg + Sufentanil 1ug/kg+ Flurbiprofen Axetil 200mg The intravenous analgesic pump in each group was supplemented with normal saline and matched to 100 ml, the background infusion rate is 2ml/h, the Self-controlled intravenous analgesia pressing once dose is 1ml, the locking time is 20min, and the analgesia lasted until 48h after surgery.
  Interventions: Drug: Esketamine 0.4mg/kg
- Esketamine experimental group (E0.6) (Experimental): Postoperative intravenous analgesia pump formula：Esketamine 0.6mg/kg + Sufentanil 1ug/kg+ Flurbiprofen Axetil 200mg The intravenous analgesic pump in each group was supplemented with normal saline and matched to 100 ml, the background infusion rate is 2ml/h, the Self-controlled intravenous analgesia pressing once dose is 1ml, the locking time is 20min, and the analgesia lasted until 48h after surgery.
  Interventions: Drug: Esketamine 0.6mg/kg
- Esketamine experimental group (E0.8) (Experimental): Postoperative intravenous analgesia pump formula：Esketamine 0.8mg/kg + Sufentanil 1ug/kg+ Flurbiprofen Axetil 200mg The intravenous analgesic pump in each group was supplemented with normal saline and matched to 100 ml, the background infusion rate is 2ml/h, the Self-controlled intravenous analgesia pressing once dose is 1ml, the locking time is 20min, and the analgesia lasted until 48h after surgery.
  Interventions: Drug: Esketamine 0.8mg/kg

INTERVENTIONS:
Drug: Esketamine is not added — Postoperative intravenous analgesia pump formula：Sufentanil 1ug/kg+ Flurbiprofen Axetil 200mg
  Arms: The control group （Esketamine is not added）
Drug: Esketamine 0.2mg/kg — Postoperative intravenous analgesia pump formula：Esketamine 0.2mg/kg + Sufentanil 1ug/kg+ Flurbiprofen Axetil 200mg.
  Arms: Esketamine experimental group(E0.2)
Drug: Esketamine 0.4mg/kg — Postoperative intravenous analgesia pump formula：Esketamine 0.4mg/kg + Sufentanil 1ug/kg+ Flurbiprofen Axetil 200ml.
  Arms: Esketamine experimental group (E0.4)
Drug: Esketamine 0.6mg/kg — Postoperative intravenous analgesia pump formula：Esketamine 0.6mg/kg + Sufentanil 1ug/kg+ Flurbiprofen Axetil 200mg.
  Arms: Esketamine experimental group (E0.6)
Drug: Esketamine 0.8mg/kg — Postoperative intravenous analgesia pump formula：Esketamine 0.8mg/kg + Sufentanil 1ug/kg+ Flurbiprofen Axetil 200mg.
  Arms: Esketamine experimental group (E0.8)

SUMMARY:
Different concentrations of Esketamine were used after cesarean section. Through the evaluation of postoperative psychological status and analgesic effect, the optimal dosage of Esketamine to exert the effects of depression and analgesia was analyzed.

DETAILED DESCRIPTION:
A total of 500 cases of pregnant women undergoing cesarean section under spinal anesthesia in Qinghai Red Cross Hospital from February 2022 to September 2022 were selected. General information of the patients were recorded, such as age, height, weight, BMI, nationality, education level, previous history, surgical history, allergy history, spouse status, fertility history and drug use status, and ASA classification was performed. Preliminarily determine whether it meets the inclusion and exclusion criteria. If it can be included in the study, the purpose, method and possible complications of the study should be fully explained to the patients and their families, as well as the significance and value of the study. Informed consent should be signed after the informed consent of the patients and their families. Patients were divided into 5 groups (n=100) according to random number method, including control group (GROUP C) and different concentrations of Esketamine dose group (group E0.2, group E0.4, group E0.6, group E0.8).

Before surgery, the puerpera were fasted for 8 hours and abstained from drinking for 4 hours. After entering the operating room, ECG monitoring and continuous oxygen inhalation by mask (2.0-3.0 L/min) were performed, and the upper limb vein channels were opened. Subarachnoid puncture was performed in L2-3 or L3-4 gaps. After the cerebrospinal fluid flows out, give 0.5% ropivacaine 10-12mg. After the subarachnoid block was successful, the epidural catheter was indurated for 4cm. The supine position was restored, and when necessary, the pregnant women were changed 30° to the left, and the supine hypotension syndrome occurred (SBP≤90mmHg or decrease ≥mmHg), 1-2mg methoxide was injected intravenously. The operation was started after the level of anesthesia was satisfied (maintain anesthesia level<T6). Postoperative intravenous controlled analgesia (PCIA). The formula of PCIA in different groups.The unified total amount of PCIA is 100mL, the background infusion rate is 2mL /h, the PCA dose is 1ml, the locking time is 20min, and the analgesia lasted until 48h after surgery.

Using SPSS26.0 statistical software. The measurement data is expressed as x±s, the comparison between groups is performed by one-way analysis of variance, the further pairwise comparison is performed by t test, and the comparison of different time points within the group is performed by repeated measures analysis of variance; the comparison of count data is performed by the chi-square test. P<0.05 indicates that the difference is statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. All participating patients signed an informed consent form;
2. Age 25-35 years old;
3. BMI≤35kg/m2;
4. ASA classification I or II;
5. Ultrasound showed a single pregnancy in the uterus Fetus, placental maturity grade Ⅱ+

Exclusion Criteria:

1. Unable or unwilling to sign the consent form, or unable to follow the research procedures;
2. History of thyroid disease;
3. A history of local anesthetic allergy;
4. A history of addiction or abuse to opioids and ketamine;
5. Preoperative mental illness; severe eclampsia;
6. Abnormal ECG, hypertension and severe heart Medical history
7. There are other contraindications to the use of esketamine

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-02-20 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Edinburgh Postpartum Depression Scale (EPDS) score | The Edinburgh Postpartum Depression Scale (EPDS) score was performed day 42 after surgery
  The Edinburgh Postpartum Depression Scale includes 10 items. According to the severity of symptoms, each item is divided into 4 levels (0, 1, 2, 3). The patient may be depressed when the total score is 10-12 points, and postpartum depression can be diagnosed when the total score is greater than 13 points.

SECONDARY OUTCOMES:
short-form of McGill Pain Questionnaire (SF-MPQ) | 6hours(T0), 12hours (T1), 24hours (T2), 48hours (T3) after operation
  The SF-MPQ consisted of 11 sensory and 4 affective descriptors for pain. All descriptors are used 0~3 to indicate the different degrees of none, light, medium and heavy respectively
Visual analog scale (VAS) for pain | 6hours (T0), 12hours(T1), 24hours (T2), 48hours (T3) after operation
  Patients were asked to circle a number that best represented their pain level using a scale of 0-10, with 0 being no pain and 10 being most severe. 0: painless; 1-3: Mild pain; 4-6: Moderate pain; 7-10: Severe pain

OTHER OUTCOMES:
The occurrence of adverse reactions | Within 48 hours after surgery
  Include hallucinations, vomiting, dizziness, and drowsiness

CONTACTS AND LOCATIONS:
Overall Officials: Wang Xuejun, director, Study Director — Department of Anesthesiology, Qinghai Red Cross Hospital

IPD SHARING:
Plan to Share IPD: Yes
Participants' basic information, depression and analgesia scores after esketamine use, and incidence of adverse reactions were shared
Supporting Information: Study Protocol, SAP, CSR
Time Frame: As of December 2025
Access Criteria: All the people

REFERENCES:
- [Background] Suppa E, Valente A, Catarci S, Zanfini BA, Draisci G. A study of low-dose S-ketamine infusion as "preventive" pain treatment for cesarean section with spinal anesthesia: benefits and side effects. Minerva Anestesiol. 2012 Jul;78(7):774-81. Epub 2012 Feb 29. PMID 22374377
- [Background] Krystal JH, Charney DS, Duman RS. A New Rapid-Acting Antidepressant. Cell. 2020 Apr 2;181(1):7. doi: 10.1016/j.cell.2020.02.033. PMID 32243798
- [Background] Singh JB, Fedgchin M, Daly E, Xi L, Melman C, De Bruecker G, Tadic A, Sienaert P, Wiegand F, Manji H, Drevets WC, Van Nueten L. Intravenous Esketamine in Adult Treatment-Resistant Depression: A Double-Blind, Double-Randomization, Placebo-Controlled Study. Biol Psychiatry. 2016 Sep 15;80(6):424-431. doi: 10.1016/j.biopsych.2015.10.018. Epub 2015 Nov 3. PMID 26707087
- [Result] O'Hara MW, McCabe JE. Postpartum depression: current status and future directions. Annu Rev Clin Psychol. 2013;9:379-407. doi: 10.1146/annurev-clinpsy-050212-185612. Epub 2013 Feb 1. PMID 23394227